CLINICAL TRIAL: NCT05154110
Title: Comparison of Static Stretching on Whole Body Vibration and Strength Training for Improving and Maintaining Hamstring Range of Motion
Brief Title: Comparison of Two Techniques for Maintaining Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Seyyada Tahniat Ali, Lecturer/Clinical instructor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FRC-BUMDC 21/ 2021
Record Dates: First submitted 2021-11-04; First posted 2021-12-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: Stretching; flexibility techniques; muscle extensibility
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strength training group (Experimental): the group will receive strength training
  Interventions: Other: strength training
- whole body vibration stretching group (Experimental): the group will receive stretching on whole-body vibration
  Interventions: Other: stretching on whole body vibration

INTERVENTIONS:
Other: stretching on whole body vibration — SSubjects will be refrained from maximum-effort or new routines for exercise the day before each treatment.Static stretching of hamstring on whole body vibration will include Pre- and post-test active and passive ROM for the both legs, with subjects first undergoing a 5-minute warm-up on a stationary bicycle. The traditional static stretch consisted of a supine active knee extension on whole body vibration (WBV) at 30 Hz at the "high" amplitude setting will be performed. The stretch will be held at the point of the onset of discomfort 3 times each for 30 seconds, with a 20-second rest period between each stretch. Participants will stretch for 4 days per week for 4 weeks. Active hamstring ROM will be measured via active knee extension using a goniometer with the leg in 90° of hip flexion, with the opposite leg extended. Passive ROM will be measured via clinician-assist ted knee extension with the leg in 90° of hip flexion.
  Arms: whole body vibration stretching group
Other: strength training — In second group, strength training will be done for 4 days per week for 4 days. Subjects will have 5 minutes warm up. In 1st week, the protocol will be Nordic hamstring curl (NHC) with bend (3 sets of 8 reps), Prone hamstrings curl (4 sets of 12 reps/leg), Physio-ball leg curl (3 sets of 8 reps), Glute bridge (2 sets of 50 s/leg). In 2nd to 4th week, the protocol will be NHC with bend (3 sets of 12 reps) Prone hamstrings curl (3 sets of 14 reps/leg) Physio-ball leg curl (3 sets of 10 reps) Glute bridge (2 sets of 50 s/leg). There will be 30 seconds rest between each set and 1 minute rest between each exercise . Pre and post AROM and PROM will be measured. Active hamstring ROM will be measured via active knee extension using a goniometer with the leg in 90° of hip flexion, with the opposite leg extended. Passive ROM will be measured via clinician-assisted knee extension with the leg in 90° of hip flexion.
  Arms: strength training group

SUMMARY:
Flexibility is a measurable physical capacity considered a key component of physical fitness. Poor flexibility is usually attributed to excessive tension exerted by the antagonist muscles of the movement and supported by weak scientific evidence, static stretching is considered as the most effective intervention in the promotion of muscle extensibility, in attempting to improve mobility.

DETAILED DESCRIPTION:
Flexibility is a measurable physical capacity considered as a key component of physical fitness thereby contributing to the health and performance of joints and the musculoskeletal system. In recent years, there has been increasing evidence that muscle weakness is a major factor behind reduced mobility. Consequently, training muscle contractility is likely to improve mobility . Regardless of terminology and of the quality of supporting evidence, stretching emerges as an intervention that elongates the tissues in attempting to improve mobility . Shortening lengthens the tissue on two out of three axes, while stretching only lengthens the tissue on one axis out of three . All training, including movement, is, by definition, training of shortening and stretching cycles (SSCs). Ergo, resistance training is also, inherently, one way to elongate . Strength training is an active, voluntary, dynamic form of stretching. Indeed, strength training is dynamic stretching. Often, strength training is performed against external resistances, but this is not mandatory. Moreover, strength training has been shown to improve mobility in sedentary adults , .

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age between 18-25
* Recreationally active individuals (all kind of sports, gym, and outdoor leisure activities)

Exclusion Criteria:

* Individuals with any physiological or pathological problem
* Older age individuals
* Individuals that had hamstring injury in past 6 months
* Individuals that had quadriceps injury in past 6 months
* Individuals that had any lower limb injury in past 6 months
* Individuals involved in any other studies.
* Individuals involved in other WBV related study.
* Sedentary lifestyle individuals

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
change in hamstring range of motion | measurements will be recoded at baseline and end of 4th week
  pre and post-change in hamstring range of motion will be assessed using a universal goniometer
maintenance of change in hamstring range of motion | measurements will be recorded after 15 days of protocol termination
  hamstring range of motion will be reassessed after 15 days using a universal goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Seyyada T Ali, Principal Investigator — bahria university medical and dental college
Locations (1):
- Seyyada Tahniat Ali, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haff, G. (2006). Roundtable Discussion: Flexibility Training. Strength and Conditioning Journal, 28(2).
- [Background] Kay AD, Blazevich AJ. Effect of acute static stretch on maximal muscle performance: a systematic review. Med Sci Sports Exerc. 2012 Jan;44(1):154-64. doi: 10.1249/MSS.0b013e318225cb27. PMID 21659901
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Result] Wan X, Li S, Best TM, Liu H, Li H, Yu B. Effects of flexibility and strength training on peak hamstring musculotendinous strains during sprinting. J Sport Health Sci. 2021 Mar;10(2):222-229. doi: 10.1016/j.jshs.2020.08.001. Epub 2020 Aug 11. PMID 32795623
- [Result] Bourne AE. Stretching with whole body vibration versus traditional static stretches to increase acute hamstring range of motion.
- [Result] Kokkonen J, Nelson AG, Tarawhiti T, Buckingham P, Winchester JB. Early-phase resistance training strength gains in novice lifters are enhanced by doing static stretching. J Strength Cond Res. 2010 Feb;24(2):502-6. doi: 10.1519/JSC.0b013e3181c06ca0. PMID 20124795